CLINICAL TRIAL: NCT00146276
Title: Adjuvant vs. Progression-Triggered Treatment With Gemcitabine After Radical Cystectomy for Locally Advanced Transitional Cell Carcinoma of the Bladder in Patients Not Suitable for Cisplatin-Based Chemotherapy - A Phase 3 Study
Brief Title: Adjuvant Versus Progression-Triggered Gemcitabine Monotherapy for Locally Advanced Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association of Urologic Oncology (AUO) (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9E-MC-S062; AB 22/00
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2005-09

CONDITIONS: Bladder Cancer; Carcinoma, Transitional Cell
Keywords: bladder cancer; cystectomy; gemcitabine; adjuvant chemotherapy; locally advanced bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine

SUMMARY:
Primary Objective:

* To analyse time to tumor progression in patients cystectomized for locally advanced transitional cell carcinoma (TCC) of the bladder, who are not suitable for cisplatin-based chemotherapy (i.e. postoperative reduced renal function, advanced age). Patients are randomized to receive either adjuvant gemcitabine immediately after radical operation (treatment arm A) or no treatment (control arm B). Patients in the control arm are to be treated with gemcitabine as soon as tumor progression becomes evident clinically and/or radiologically.

Secondary Objectives:

The secondary objectives of this study are:

* Estimation of time-specific survival probabilities irrespective of causes of death.
* Assessment of toxicity and tolerability of gemcitabine
* Description of survival experience of patients in the control arm beyond the time of initiating chemotherapy.
* Assessment of quality of life (European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-C30).

Study Design:

This is an open-label, prospective, multicenter, randomized, controlled phase 3 two-arm study using gemcitabine as a single agent in chemonaive cystectomy patients with locally advanced TCC of the bladder in an adjuvant setting. The patients will receive the following treatment:

Arm A (treatment): gemcitabine 1250 mg/m2 intravenously once a week for 2 weeks (days 1 and 8) followed by 1-week rest period. Repeat cycle on day 22. Maximum of 6 cycles. Begin treatment until 3 months after radical operation (within first 6 weeks is recommended).

Arm B (control): No immediate post-surgery treatment. Watchful waiting; treatment only conditionally in case of progression with gemcitabine (dose and schedule as in arm A).

DETAILED DESCRIPTION:
Primary Objective:

* To analyse time to tumor progression in patients cystectomized for locally advanced TCC of the bladder, who are not suitable for cisplatin-based chemotherapy (i.e. postoperative reduced renal function, advanced age). Patients are randomized to receive either adjuvant Gemcitabine immediately after radical operation (treatment arm A) or no treatment (control arm B). Patients in the control arm are to be treated with Gemcitabine as soon as tumor progression becomes evident clinically and/or radiologically.

Secondary Objectives:

The secondary objectives of this study are:

* Estimation of time-specific survival probabilities irrespective of causes of death.
* Assessment of toxicity and tolerability of Gemcitabine
* Description of survival experience of patients in the control arm beyond the time of initiating chemotherapy.
* Assessment of quality of life (EORTC QLQ-C30).

Study Design:

This is an open-label, prospective, multicenter, randomized, controlled phase 3 two-arm study using Gemcitabine as a single agent in chemonaive cystectomy patients with locally advanced TCC of the bladder in an adjuvant setting. The patients will receive the following treatment:

Arm A (treatment): Gemcitabine 1250 mg/m2 intravenously once a week for 2 weeks (days 1 and 8) followed by 1-week rest period. Repeat cycle on day 22. Maximum of 6 cycles. Begin treatment until 3 months after radical operation (within first 6 weeks is recommended).

Arm B (control): No immediate post-surgery treatment. Watchful waiting; treatment only conditionally in case of progression with Gemcitabine (dose and schedule as in arm A).

ELIGIBILITY:
Inclusion Criteria:

* Status after radical cystectomy for transitional cell carcinoma of the bladder, stages pT3a, pT3b, pT4a and/or pN1, pN2 (but no more than 5 lymph nodes positive for tumor) [International Union Against Cancer (UICC) criteria, 1997]. Transitional cell carcinoma may be with or without squamous cell carcinoma and/or adenocarcinoma components. Complete tumor removal by radical operation has to be established macroscopically and microscopically (R0 resection).
* Patients regarded as inappropriate for cisplatin-based chemotherapy (i.e. impaired renal function with at least 30 ml/min calculated creatinine clearance and serum-creatinine less than 3.0 mg/dl, age > 70) are eligible for study enrollment [calculation of creatinine clearance according to Cockcroft and Gault formula]. Decision left to the investigator's discretion.
* Patient has no prior history of systemic chemotherapy regimens. Previous local intravesical adjuvant chemotherapy or immunotherapy is allowed.
* Prior radiation therapy is allowed if it has been completed at least 12 weeks before enrollment into the study and the patient has recovered from all toxic effects.
* Performance status of 60 or higher on the Karnofsky Scale.
* Patient compliance, mental state, and geographic proximity allow adequate followup
* Adequate bone marrow reserve: white blood cell (WBC) count >= 3.5 x 10^9/L, platelets >= 100 x 10^9/L, and hemoglobin >= 10 g/dL (or >= 6.2 mmol/L or >= 100 g/L).
* Adequate liver function with bilirubin < 1.25 times above upper limit of normal range; alanine transaminase (ALT) or aspartate transaminase (AST) < 2.5 times normal upper limit.
* Males or females at least 18 years of age who are considered fit for gemcitabine chemotherapy.
* Signed informed consent by the patient.

Exclusion Criteria:

* Tumor was not completely removed (visible tumor or enlarged lymph nodes left or positive margins microscopically-R1 or R2 resection)
* Patient has a distant metastasis or metastases.
* Tumor stage pT4b or more than 5 locoregional lymph nodes are positive for tumor.
* Adeno- and/or squamous cell carcinoma of the bladder without transitional cell carcinoma component (different responses to chemotherapy).
* Time interval between radical cystectomy and the first day of chemotherapy exceeds 3 months for patients enrolled in the treatment arm.
* Serum creatinine >= 3.0 mg/dl (>= 265 mmol/l)
* Active infection (at the discretion of the investigator) .
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Patients with a history of prior malignancy other than basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or incidental carcinoma of the prostate must be clinically free of disease for at least 5 years prior to study entry.
* Use of any investigational agent in the month before enrollment into the study.
* White blood cell (WBC) count < 3.5 x 10^9/L or platelets < 100 x 10^9/L or hemoglobin < 10 g/dL (or < 6.2 mmol/L or < 100 g/L).
* Bilirubin >= 1.25 times above upper limit of normal range; alanine transaminase (ALT) or aspartate transaminase (AST) >= 2.5 times upper limit of normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178
Dates: Start 2000-07

PRIMARY OUTCOMES:
progression-free survival

SECONDARY OUTCOMES:
overall survival
toxicity and tolerability of gemcitabine
quality of life (EORTC QLQ-C30, version 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stöckle, MD, Principal Investigator — Dept of Urology, Saarland University
Locations (1):
- Saarland University, Homburg/Saar, Saarland, Germany

REFERENCES:
- See also: see "Aktivierte Studien/Blase" — http://www.auo-online.de